CLINICAL TRIAL: NCT02815410
Title: The Prospective Trial for Validation of the Role of Levetiracetam as a Sensitizer of Temozolomide in the Treatment of Newly Diagnosed Glioblastoma Patients
Brief Title: Validation of the Role of Levetiracetam for Newly Diagnosed GBM Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chae-Yong Kim, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: cykim
Record Dates: First submitted 2016-06-14; First posted 2016-06-28 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Glioblastoma Multiforme
Keywords: Glioblastoma Multiforme; Levetiracetam; Temozolomide; Survival outcome
MeSH Terms: conditions — Glioblastoma | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Levetiracetam (Other): Newly diagnosed histologically proven supratentorial glioblastoma patients received levetiracetam during and after their CCRT
  Interventions: Drug: levetiracetam

INTERVENTIONS:
Drug: levetiracetam — Patients in this group are with newly diagnosed glioblastoma patients who are supposed to be treated with concurrent chemoradiotherapy (CCRT) and adjuvant chemotherapy with temozolomide (TMZ). Patients ( intervention Group) will be given levetiracetam (LEV) from the beginning of treatment till after the adjuvant chemotherapy with TMZ is over.
  Other Names: keppra®

SUMMARY:
Prospective, open-labeled, multicenter cohort trial for validation of the role of levetiracetam as a sensitizer of temozolomide in the treatment of newly diagnosed glioblastoma patients.

DETAILED DESCRIPTION:
I. Objectives

<Primary Endpoint>

6 months progression-free survival (6m-PFS)

<Secondary Endpoint>

1. Overall survival
2. Safety (adverse events)
3. Quality of life using EORTC module,
4. Cognitive function using NOPT module of our institution

<Explorative Endpoint>

Genetic biomarker for predicting prognosis

1. Methylation status of MGMT promoter
2. IDH mutation
3. TERT mutation / ATRX status

II. Hypothesis

1.Proof of concept

* With using of levetiracetam, there will be an improved survival with chemoradiotherapy with temozolomide compared to the group without using levetiracetam. (superiority) 2. Safety
* It will be tolerable in this concept. 3. Genetic biomarker
* Methylation status of MGMT, IDH1 mutation, TERT mutation, and ATRX status will prove to be valid molecular markers of prognostic significance in newly diagnosed glioblastoma treated with the combination of levetiracetam.

III. Study Design/Clinical Plan

1. Group I (prospective)

   * Patients in this group are with newly diagnosed glioblastoma patients who are supposed to be treated with concurrent chemoradiotherapy (CCRT) and adjuvant chemotherapy with temozolomide (TMZ). Patients in Group I will be given levetiracetam (LEV) from the beginning of treatment till after the adjuvant chemotherapy with TMZ is over.
2. Group II (historical group; using data base from KSNO multicenter study group)

IV. Treatment

1. Levetiracetam: started with 250mg bid and is increased up to 500mg bid in perioperative period. During the 2 days of peri-operation, it is administered in intravenous form mixed in 150ml of normal saline. After immediate postoperative period, 500~1500mg bid is administered in per oral form according to patient's clinical condition. During the period of adjuvant chemotherapy with temozolomide, the dose not less than 500mg is administered unless there are serious side effects of levetiracetam.
2. Temozolomide based standard treatment: CCRT with temozolomide followed by 6cycles of adjuvant temozolomide RT with daily temozolomide (75 mg/m2/day, 7 days/week) from the first to the last day of radiotherapy), followed by six cycles of adjuvant temozolomide (150 to 200 mg/m2 for 5 days during each 28-day cycle).

V. Evaluation

MR scans were performed before the first adjuvant treatment cycle and then every 3 months during the first year, and every 4 months during the second year. Radiographic response is determined in comparison to the tumor measurement obtained at pretreatment baseline measurements as a reference and is categorized into four groups using new criteria proposed by the Response Assessment in Neuro-Oncology (RANO) working group.

VI. Statistical Plans

Total sample size: 73 The size of sample is considered by assessment of PFS. The number of event and statistical power was calculated on assumption of exponential distribution of the 7 months median PFS in the control group and 12 months median PFS in the treatment group.

The expected sample size provides 80% of test power that can perceive 1.7 of hazard ration with 0.05 of type I error in comparative analysis of PFS at the time of 12 months of registering period (in equal entry pattern) and at 6 months of follow up period. Basis on this assumption, it is expected that 73 patients are needed in the treatment group, and 74 patients in the control group.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed histologically proven supratentorial glioblastoma (World Health Organization [WHO] Grade IV). The histological diagnosis must be obtained from a neurosurgical resection or biopsy of a tumor including an open biopsy or stereotactic biopsy.
2. Age 20 -76 years
3. Eastern Cooperative Oncology Group performance status (ECOG PS) of 0-2
4. Meets 1 of the following RPA classifications:

   4-1. Class III (Age <50 years and ECOG PS 0) 4-2. Class IV (meeting one of the following criteria: a) Age <50 years and ECOG PS 1 or b) Age ≥50 years, underwent prior partial or total tumor resection, MMSE ≥27) 4-3. Class V (meeting one of the following criteria: a) Age ≥50 years and underwent prior partial or total tumor resection, MMSE <27 or b) Age ≥50 years and underwent prior tumor biopsy only)
5. Adequate hematologic, renal, and hepatic function:

   ANC > 1,500/uL Platelet > 100,000/uL Serum creatinine <1.7mg/dL Bilirubin level < 2.0 mg/dL AST/ALT < 2.5 x upper limit of normal range of each institution
6. Written informed consent

Exclusion Criteria:

1. Prior chemotherapy within last 5 years
2. Prior radiotherapy of the head and neck area
3. Receiving concurrent investigational agents or has received an investigational agent within 30 days prior to randomization
4. Planned surgery for other diseases (e.g. dental extraction)
5. History of malignancy. Subjects with curatively treated cervical carcinoma in situ or basal cell carcinoma of the skin, or subjects who have been free of other malignancies for 5 years are eligible for this study
6. Pregnant or lactating women
7. Subject who disagree to follow acceptable methods of contraception
8. Concurrent illness including unstable heart disease despite appropriate treatment, history of myocardial infarction within 6 months, serious neurological or psychological disease, and uncontrolled infection

Ages: 20 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2016-07; Primary Completion 2019-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
6 months Progression free survival | from the first operation to following 6 months

SECONDARY OUTCOMES:
Overall survival | from the first operation to following 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Chae-Yong Kim, PhD, Principal Investigator — Seoul National University Bundang Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim YH, Kim T, Joo JD, Han JH, Kim YJ, Kim IA, Yun CH, Kim CY. Survival benefit of levetiracetam in patients treated with concomitant chemoradiotherapy and adjuvant chemotherapy with temozolomide for glioblastoma multiforme. Cancer. 2015 Sep 1;121(17):2926-32. doi: 10.1002/cncr.29439. Epub 2015 May 14. PMID 25975354
- [Background] Guthrie GD, Eljamel S. Impact of particular antiepileptic drugs on the survival of patients with glioblastoma multiforme. J Neurosurg. 2013 Apr;118(4):859-65. doi: 10.3171/2012.10.JNS12169. Epub 2012 Nov 23. PMID 23176328
- [Background] Kerkhof M, Dielemans JC, van Breemen MS, Zwinkels H, Walchenbach R, Taphoorn MJ, Vecht CJ. Effect of valproic acid on seizure control and on survival in patients with glioblastoma multiforme. Neuro Oncol. 2013 Jul;15(7):961-7. doi: 10.1093/neuonc/not057. Epub 2013 May 16. PMID 23680820
- [Derived] Hwang K, Kim J, Kang SG, Jung TY, Kim JH, Kim SH, Kang SH, Hong YK, Kim TM, Kim YJ, Choi BS, Chang JH, Kim CY. Levetiracetam as a sensitizer of concurrent chemoradiotherapy in newly diagnosed glioblastoma: An open-label phase 2 study. Cancer Med. 2022 Jan;11(2):371-379. doi: 10.1002/cam4.4454. Epub 2021 Nov 30. PMID 34845868